CLINICAL TRIAL: NCT02451722
Title: Evaluation of Pressure Distribution of Kyboot Shoes in Comparison to Other Foot Wear in Diabetic Patients and in Healthy Subjects
Brief Title: Evaluation of Pressure Distribution of Kyboot Shoes in Comparison to Other Foot Wear
Acronym: Kyboot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Kybun AG (Unknown)
Responsible Party: Principal Investigator, Dr. Itzhak Siev-Ner, Head of Orthopedic Rehabilitation department, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHEBA-2053-15-SMC
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus Type 2; Sensory Neuropathy; Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy subjects (Active Comparator): Kyboot shoes will be administered to the healthy subjects.
  Pressure distribution and gait parameters will be recorded in comparison with their normal footwear.
  Interventions: Device: Kyboot shoes
- Diabetic patients (Active Comparator): Kyboot shoes will be administered to the diabetic patients.
  Pressure distribution and gait parameters will be recorded in comparison with their normal footwear.
  Interventions: Device: Kyboot shoes

INTERVENTIONS:
Device: Kyboot shoes — The Kyboot shoe - construction is based on a soft, supple air cushioned sole. The honeycomb air structure of the kyBoot sole creates an air cushion between your foot and the ground, with one fifth of the volume of air being pumped into the foot area at every step. This design could offer a better distribution of pressure
  Other Names: Kybun shoe

SUMMARY:
Comparison and evaluation of pressure distribution, gait pattern, changes in the movement of the center of pressure, shock absorbing capabilities and comfort of wear using KyBoot shoes versus normal foot wear in diabetic and healthy subjects.

DETAILED DESCRIPTION:
Every 30 seconds a limb is lost somewhere in the world as a consequence of diabetes. These amputations are preceded by a foot ulcer in 84% of cases. Therefore, prevention of ulceration is of utmost importance.

Approximately one-half of all diabetic foot ulcers occur on the plantar foot surface and are mainly caused by elevated levels of mechanical pressure acting on the foot during ambulation in the presence of lost protective foot sensation from peripheral neuropathy.

Therefore, to reduce risk of ulceration, relief of mechanical pressure (also called offloading) is indicated.

Currently therapeutic footwear is provided by the Health maintenance organizations (HMO's) to diabetic patients that are at risk of developing foot ulcers.

Ideal footwear for a diabetic patient decreases weight-bearing pressure and shear forces applied to the skin of the foot by distributing the acting forces more evenly.

With the growth in the health and fitness industry, sports footwear has shown technological advances and diversification.

The introduction of the KyBoot shoe is an example of this diversification. The Kybun company based their shoe on the experience of walking on soft, muddy rice fields in Korea.

The Kyboot construction is based on a soft, supple air cushioned sole. The honeycomb air structure of the kyBoot sole creates an air cushion between your foot and the ground, with one fifth of the volume of air being pumped into the foot area at every step. This design could offer a better distribution of pressure.

Therefore, in this study we would like to compare the pressure distribution, changes in the movement of the center of pressure and shock absorbing capabilities of the KyBoot in comparison with normal shoes.

Study goals:

Comparison and evaluation of pressure distribution, gait pattern, changes in the movement of the center of pressure, shock absorbing capabilities and comfort of wear using KyBoot shoes versus normal foot wear in diabetic and healthy subjects.

ELIGIBILITY:
Inclusion Criteria: ( for the group of diabetic patients)

* Signing of informed consent
* Diabetes mellitus Type 2
* No major foot deformations necessitating fitting of personalized foot wear
* Absence of diabetic foot ulcers and existence of sensory neuropathy confirmed by a physician
* Intact cognitive function
* Normal Gait

Exclusion Criteria:

* An orthopedic or rheumatic disease that negatively influences range of motion, strength, gait or balance
* Neurological diseases that influence proprioception , strength, balance, cognitive function / understanding, sight: Cerebro-vascular accident, Dementia, Spinal Cord injury, Head injury, Parkinson etc.
* Injury or disease that can influence normal gait
* Need for assistive devices : Crutches, cane, walker
* Dialysis Treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Reduction of Peak Pressure | 1 day
  The pressure distribution will be measured by in-sole pressure sensors.

SECONDARY OUTCOMES:
Comfort of wear | 1 Day
  Comfort of wear will be evaluated with the help of a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Itzhak Siev-Ner, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Orthopedic Rehabilitation out-patient clinic, Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Boulton AJ, Vileikyte L, Ragnarson-Tennvall G, Apelqvist J. The global burden of diabetic foot disease. Lancet. 2005 Nov 12;366(9498):1719-24. doi: 10.1016/S0140-6736(05)67698-2. PMID 16291066
- [Background] Pecoraro RE, Reiber GE, Burgess EM. Pathways to diabetic limb amputation. Basis for prevention. Diabetes Care. 1990 May;13(5):513-21. doi: 10.2337/diacare.13.5.513. PMID 2351029
- [Background] Pham H, Armstrong DG, Harvey C, Harkless LB, Giurini JM, Veves A. Screening techniques to identify people at high risk for diabetic foot ulceration: a prospective multicenter trial. Diabetes Care. 2000 May;23(5):606-11. doi: 10.2337/diacare.23.5.606. PMID 10834417
- [Background] Prompers L, Huijberts M, Apelqvist J, Jude E, Piaggesi A, Bakker K, Edmonds M, Holstein P, Jirkovska A, Mauricio D, Ragnarson Tennvall G, Reike H, Spraul M, Uccioli L, Urbancic V, Van Acker K, van Baal J, van Merode F, Schaper N. High prevalence of ischaemia, infection and serious comorbidity in patients with diabetic foot disease in Europe. Baseline results from the Eurodiale study. Diabetologia. 2007 Jan;50(1):18-25. doi: 10.1007/s00125-006-0491-1. Epub 2006 Nov 9. PMID 17093942
- [Background] Bus SA, Valk GD, van Deursen RW, Armstrong DG, Caravaggi C, Hlavacek P, Bakker K, Cavanagh PR. The effectiveness of footwear and offloading interventions to prevent and heal foot ulcers and reduce plantar pressure in diabetes: a systematic review. Diabetes Metab Res Rev. 2008 May-Jun;24 Suppl 1:S162-80. doi: 10.1002/dmrr.850. PMID 18442178
- See also: The company providing the Kyboot shoe — http://www.kybun.com